CLINICAL TRIAL: NCT06292169
Title: A Randomized Control Trial to Evaluate Release Versus Non-release of Pectoralis Minor With Reverse Shoulder Arthroplasty
Brief Title: Pectoralis Minor Release Versus Non-release in RSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Eric Wagner, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007201
Record Dates: First submitted 2024-02-15; First posted 2024-03-05 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Reverse Total Shoulder Arthroplasty; Rotator Cuff Tear Arthropathy; Advanced Glenohumeral Osteoarthritis
Keywords: Reverse Total Shoulder Arthroplasty; Reverse Shoulder Arthroplasty; American Shoulder and Elbow; Range of motion; Pectoralis Minor
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Electronic random number generator Single-blinded (concealed to the study participant only, Investigator blinded not feasible)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RSA with pectoralis minor release (Experimental)
  Interventions: Procedure: Pectoralis Minor Release; Procedure: RSA
- RSA without pectoralis minor release (Active Comparator)
  Interventions: Procedure: RSA

INTERVENTIONS:
Procedure: Pectoralis Minor Release — The pectoralis minor is a muscle on the anterior chest wall attaching to the coracoid process. In the group undergoing pectoralis minor release, through the same deltopectoral incision that will not be extended or different as compared to the RSA only group, the pec minor will be exposed on the medial aspect of the coracoid at the upper part of the incision. It will be cut from its insertion on the coracoid while being careful to protect any neurovascular structures.
  Arms: RSA with pectoralis minor release
Procedure: RSA — RSA is the current Standard of Care (SOC)

SUMMARY:
The goal of this clinical trial is to assess if concomitant open pectoralis minor release would improve pain and outcomes after Reverse Shoulder Arthroplasty (RSA). The main questions it aims to answer are:

* whether releasing the pectoralis minor prophylactically could have better pain relief
* whether releasing the pectoralis minor prophylactically could have increased Range of motion (ROM) outcomes
* whether releasing the pectoralis minor prophylactically could have higher final Patient Reported Outcome Measurements (PROMs) Participants will be randomized to either undergo RSA with pectoralis minor release or RSA without pectoralis minor release.

DETAILED DESCRIPTION:
Shoulder arthroplasty has been increasing at exponential rates, particularly due to the rise of reverse shoulder arthroplasty (RSA). Postoperative complications after RSA include infection, instability, hardware component loosening, acromial and scapular spine fractures, neurologic injury, and scapular notching which can all cause pain. However, despite excluding these causes, some patients can have persistent anterior shoulder pain with poor motion.

RSA prostheses work by translating the center of rotation (COR) inferiorly and medially, which increases tension on the deltoid, which is thought to increase the deltoid's mechanical moment arm and thus its ability to abduct and flex the humerus. However, excessive lengthening may be a cause of acromial and scapular spine fractures or neurologic injury. In addition, other structures are tensioned, including the conjoint tendon (short head of the biceps brachii and coracobrachialis) and pec minor (PM). It is unclear if lengthening these muscle-tendon units has functional consequences or whether it can create an intrinsic pathology. It is therefore feasible that muscle lengthening could create tendinitis, which could lead to persistent anterior shoulder pain after RSA. In addition, excessive tension or over-activity in the PM is also known to be a cause of altered scapula biomechanics.

Good scapula biomechanics after RSA are critical to preserving an impingement-free range of motion, which is important in maximizing postoperative outcomes, implant longevity, and preventing component loosening and instability. However, it is known from the non-arthroplasty population that during repetitive movements with scapular protraction, a hyperactive or spasming PM shortens and develops contracture, leading to protracted resting scapular position and altered scapular contribution to shoulder range of motion.1 This causes altered scapular kinematics, or dyskinesia, and alters scapular accommodation to shoulder motion, a well-known feature in various shoulder pathologies. This can be a major problem after RSA when scapula accommodation is critical to ROM and function.

Due to the expendability of the pectoralis minor, its release would cause minimal functional detriment in non-pathological cases, but in cases of overactivity, release could markedly improve scapula biomechanics. This can be performed open or arthroscopically, but the concomitant open release would be straight-forward at the time of the index surgery through the same incision

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing surgery for reverse total shoulder arthroplasty
* Patients willing and able to provide informed consent

Exclusion Criteria:

* Revision arthroplasty
* Reverse shoulder arthroplasty for proximal humerus fractures
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog Scale (VAS) pain scores | Baseline, 6 months
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Study participants will be asked to rate their current level of pain by placing a mark on the line

OTHER OUTCOMES:
Visual analog Scale (VAS) pain scores | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year (each follow-up visit)
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Study participants will be asked to rate their current level of pain by placing a mark on the line
American Shoulder and Elbow Score (ASES) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year (each follow-up visit)
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points.
Subjective Shoulder Value (SSV) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year (each follow-up visit)
  Subjective Shoulder Value is study participant's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%
Change in Range of motion (ROM) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year (each follow-up visit)
  ROM is calculated in terms of angles. Lower number suggests restricted motion.
Change in Scapulohumeral Rhythm (SHR) on Digital Dynamic Radiography (DDR) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year (each follow-up visit)
  SHR is the ratio of humeral abduction over the change in scapula upward rotation during humeral abduction. This SHR will be captured on Digital Dynamic Radiography (DDR) and reported as a change in SHR before and after the interventions.
Number of complications | 1 year
  Number of complications post intervention would be measured.
Number of reoperations | 1 year
  Number of reoperations following intervention would be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wagner, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Clinic, Atlanta, Georgia
  - Emory Healthcare Orthopaedics and Spine Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No